CLINICAL TRIAL: NCT02582970
Title: An Expanded Access Program of AvastinTM (Bevacizumab) in Patients With Metastatic Cancer of the Colon or Rectum
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Chemotherapy in Participants With Metastatic Cancer of the Colon or Rectum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18436
Record Dates: First submitted 2015-10-12; First posted 2015-10-21 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Irinotecan; Oxaliplatin

ARMS (1):
- Bevacizumab + Chemotherapy (Experimental): Participants will receive IV bevacizumab at a dose of 5 milligrams per kilogram (mg/kg) every 2 weeks in combination with standard of care chemotherapy regimen (5-Fluorouracil/Irinotecan/Oxaliplatin) until disease progression or until termination of the study.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — Intravenous 5-fluorouracil based chemotherapy will be administered until disease progression or until termination of the study. The chemotherapy regimen will be at the discretion of the prescriber and will not be provided by the sponsor.
Drug: Bevacizumab — Bevacizumab will be administered IV 5 mg/kg every 2 weeks until disease progression or until termination of the study.
  Other Names: Avastin
Drug: Irinotecan — Irinotecan will be administered at the discretion of the prescriber until disease progression or until termination of the study.
Drug: Oxaliplatin — Oxaliplatin will be administered at the discretion of the prescriber until disease progression or until termination of the study.

SUMMARY:
This expanded access study will assess the efficacy and safety of intravenous (IV) bevacizumab in combination with chemotherapy regimens as first-line treatment of metastatic cancer of the colon or rectum. The anticipated median time on study treatment is approximately 10 months, and the target sample size is 40 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated metastatic colon or rectal cancer
* Scheduled to begin IV 5-fluorouracil-based chemotherapy as a first-line treatment

Exclusion Criteria:

* Prior chemotherapy for metastatic colon or rectal cancer
* Planned radiotherapy for underlying disease
* Central nervous system metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study start
* Treatment with any investigational drug, or participation in another investigational study, within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (5):
- Taiwan (5):
  - Chai Yi
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Chemotherapy: Participants received bevacizumab at a dose of 5 milligrams per kilogram (mg/kg) every 2 weeks (q2w) in combination with standard chemotherapy regimen (5-Fluorouracil/Irinotecan/Oxaliplatin) until disease progression or until termination of the study.
Period: Overall Study
Arm/Group | Bevacizumab + Chemotherapy
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants receiving at least one dose of study drug.
Groups:
- Bevacizumab + Chemotherapy: Participants received bevacizumab at a dose of 5 mg/kg q2w in combination with standard chemotherapy regimen (5-Fluorouracil/Irinotecan/Oxaliplatin) until disease progression or until termination of the study.
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was any untoward medical occurrence attributed to study drug in a participant who received study drug.
Time Frame: Baseline up to approximately 3 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
percentage of participants | 100

2. Secondary Outcome: Percentage of Participants Who Died
Time Frame: Baseline up to approximately 3 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
percentage of participants | 62.5

3. Secondary Outcome: Duration of Survival
Description: Duration of survival was defined as the time period from the start of first line therapy to death. Duration of survival was estimated using Kaplan-Meier analysis.
Time Frame: Baseline up to approximately 3 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
months | 23.8 [13.7 to 27.2]

4. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression was defined as at least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions, or evidence of clinical progression and unequivocal progression of existing non-target lesions (TL).
Time Frame: Baseline up to approximately 3 years
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
percentage of participants | 85.0

5. Secondary Outcome: Progression-Free Survival Time
Description: Progression-free survival was defined as the duration from the date of starting first-line therapy to the date of documented disease progression or death from any cause. Disease progression was defined as at least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions, or evidence of clinical progression and unequivocal progression of existing non-TL. Progression-free survival was estimated using Kaplan-Meier analysis.
Time Frame: Baseline up to approximately 3 years
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
months | 12.2 [9.4 to 15.9]

6. Secondary Outcome: Number of Participants With Best Overall Response
Description: The best overall response was defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Progressive disease (PD): at least a 20% increase in the disease measurement, taking as reference the smallest disease measurement recorded since the start of treatment, or the appearance of one or more new lesions, or evidence of clinical progression and unequivocal progression of existing non-TL. Complete response (CR): disappearance of all TL and non-TL. If immunocytology was available, no disease was to be detected by that methodology. Partial response (PR): at least a 30% decrease in the disease measurement, taking as reference the disease measurement done to confirm measurable disease at study entry. Stable disease (SD): neither sufficient shrinkage to qualify for PR or increase to qualify for PD.
Time Frame: Baseline up to approximately 3 years
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 40
participants
  CR | 2
  PR | 19
  PD | 8
  SD | 9
  Missing | 2

7. Secondary Outcome: Mean Direct Medical Cost for Cancer Related Medical Care Utilization
Description: Direct medical cost included cost of out-patient consultation and cost of hospitalization.
Time Frame: Baseline up to approximately 3 years
Population: ITT population. Here, number of participants analyzed = participants who were evaluable for this outcome measure. Number Analyzed = participants who were evaluable for specified categories of this outcome measure.
Measure: Mean (Standard Deviation); unit: Thousands in New Taiwan Dollar
Arm/Group | Bevacizumab + Chemotherapy
Number analyzed (Participants) | 14
Thousands in New Taiwan Dollar
  Out-Patient Consultation: number analyzed (Participants) | 13
  Out-Patient Consultation | 0.91 (0.407)
  Hospitalization | 35.9 (12.8)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 3 years
Groups:
- Bevacizumab + Chemotherapy: Participants received IV bevacizumab at a dose of 5 mg/kg q2w in combination with standard of care chemotherapy regimen until disease progression or until termination of the study.
Arm/Group | Bevacizumab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=40)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Disease progression (General disorders) | 1
Pyrexia (General disorders) | 1
Abscess (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=40)
Leukopenia (Blood and lymphatic system disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 22
Gastrointestinal disorder (Gastrointestinal disorders) | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 27
Periodontal disease (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 13
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 24
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 2
Fatigue (General disorders) | 24
Impaired healing (General disorders) | 2
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 12
Hypersensitivity (Immune system disorders) | 3
Urinary tract infection (Infections and infestations) | 3
Sensory level abnormal (Investigations) | 11
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 15
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 11
Neuropathy peripheral (Nervous system disorders) | 11
Insomnia (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 15
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Flushing (Vascular disorders) | 7
Haemorrhage (Vascular disorders) | 3
Hypertension (Vascular disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.